CLINICAL TRIAL: NCT05069961
Title: Non- Inferiority Study of Erector Spinae Plane Block Compared to Thoracic Epidural Analgesia in Multimodal Pain Management of Multiple Rib Fractures
Brief Title: Non-Inferiority Study of Erector Spinae Plane Block Compared to Thoracic Epidural in Pain Management of Rib Fractures
Acronym: SUETHE-Ribs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was closed with IRB as PI wants to design the protocol extensively.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Ross Mirman, Assistant Professor of Clinical Anesthesia, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11414
Record Dates: First submitted 2021-09-03; First posted 2021-10-06 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB Group (Active Comparator): 20ml Ropivacaine is injected near the nerves in the back and then continued using an infusion pump.
  Interventions: Procedure: ESPB
- TEA Group (Active Comparator): 5ml Bupivacaine is injected into the space around the spinal cord and then continued using an infusion pump.
  Interventions: Procedure: TEA

INTERVENTIONS:
Procedure: ESPB — Ropivacaine is injected near the nerves in the back
  Arms: ESPB Group
Procedure: TEA — Bupivacaine is injected into the space around the spinal cord.
  Arms: TEA Group

SUMMARY:
The purpose of this study is to compare 2 pain control treatments for people with 3 or more rib fractures.

DETAILED DESCRIPTION:
2.1 Primary Objective

* Compare efficacy of ESPB to TEA for MRF analgesia.

2.2 Secondary Objective

* Compare systemic opioid and non-opioid medication use in patients with ESPB and TEA.

2.3 Tertiary/Exploratory/Correlative Objectives

* Determine improvement in respiratory function in ESPB versus TEA before and after analgesia placement.
* Compare complications that occur in patients who receive ESPB versus TEA.
* Compare dermatome levels relative to catheter placement that achieve analgesia for TEA and ESPB.
* Compare differences in deep vein thrombosis (DVT) prophylaxis and incidence between ESPB and TEA.
* Differences in length of stay (LOS) for TEA versus ESPB.
* Differences in risk of delirium between TEA and ESPB.
* Differences in oxygen and ventilatory support between TEA and ESPB.
* Patient satisfaction of pain management.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Radiological evidence of 3 or more rib fractures
* Within 48 hours of admission to hospital with rib fractures
* Can actively participate by answering questions during TEA or ESPB placement
* Moderate-severe (4-10 out of 10) pain at the time of enrollment

Exclusion Criteria:

* Greater than 48 hrs since admission to the hospital with rib fractures
* Patient refusal
* Prisoner
* Infection at the site of TEA or ESPB insertion
* Allergy to local anesthetics
* Depth from skin to catheter placement target 6 or more centimeters
* Greater than 7 consecutive ribs involved on each side
* Other regional or epidural block already received
* Unable to follow commands/altered mental status
* Dementia
* Sepsis (temperature > 38 degrees Celsius & positive blood cultures)
* Elevated intracranial pressure (ICP > 12 mm Hg)
* Coagulopathy (INR > 1.4) or recent therapeutic anticoagulant use (varies with which medication the patient is on)
* Preexisting central nervous system disorders, such as multiple sclerosis
* Thrombocytopenia (Platelets <70,000)
* Spine fracture or previous back surgery
* Preload dependent states (aortic stenosis, hypertrophic obstructive cardiomyopathy)
* Aortic transection
* Hemodynamic instability (patients with MAPs <60 and/or patients requiring pressor support)
* Tattoo at sight of catheter placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
MRF pain at rest and with cough before and after TEA or ESPB placement using the pain visual analog scale (VAS) for pain in the thorax/ribs. | 24 hours after catheter placement
  Participants will be asked about their rib pain specifically during this assessment along with the maximum pain experienced and its location. VAS is used to measure pain on a scale of 1-10, with 1 being the least and 10 being the most amount of pain.
MRF pain at rest and with cough before and after TEA or ESPB placement using the pain visual analog scale (VAS) for pain in the thorax/ribs. | 72 hours after catheter placement
  Participants will be asked about their rib pain specifically during this assessment along with the maximum pain experienced and its location. VAS is used to measure pain on a scale of 1-10, with 1 being the least and 10 being the most amount of pain.

SECONDARY OUTCOMES:
Determine total systemic opioid and non-opioid medication use in patients with ESPB and TEA by reviewing patient EMR. | After patient discharge up to 7 days
  Normalize medication use by subtracting baseline opioid and non-opioid medication use for amount received while hospitalized and compare injury severity prior to analysis.

OTHER OUTCOMES:
Incentive spirometry | Baseline, pre-intervention and immediately following intervention.
  Maximum incentive spirometry volume (in mL) will be gathered.
Rate of adverse events/complications related to ESPB and TEA | Duration of hospital stay up to 7 days.
  Track adverse events/complications related to ESPB and TEA such as pneumothorax, pneumonia, infection at catheter site, DVT, pulmonary embolism, urinary retention, hypotension, spinal cord injury, systemic anesthetic toxicity, epidural hematoma, and loss of motor function.
Dermatome levels with analgesia | Immediately following infusion.
  Determine dermatome levels with analgesia using via cold sensory.
Dermatome levels with analgesia | 30 minutes after infusion.
  Determine dermatome levels with analgesia using via cold sensory.
Dermatome levels with analgesia | Once a day in the morning, after intervention. They will be checked until the catheter is removed, which will be 7 days at the longest.
  Determine dermatome levels with analgesia using via cold sensory.
Risk assessment profile (RAP) score | After patient discharge up to 7 days
  Standard trauma protocol includes all trauma inpatients getting a risk assessment profile (RAP) score. A RAP score <5 needs no additional monitoring. A RAP score >/= 5 gets anti-Xa monitoring (4 hrs after 3rd consecutive dose with goal parameters 0.2-0.4). A RAP score >/= 11 gets Anti-Xa monitoring plus weekly lower extremity dopplers ultrasound. This data will be in the EMR as it is standard protocol currently.
The time spent in the intensive care unit (ICU) | Duration of hospital stay, up to 7 days.
  Total time spent in ICU
Total length of hospital stay | Up to 7 days.
  Amount of time each subject spends in the hospital before discharge.
Confusion assessment method (CAM-ICU) | Daily during hospital stay up to 7 days.
  Scores will be charted daily and reviewed in the EMR to determine if differences in delirium are present for patients receiving TEA versus ESPB
Richmond Agitation-Sedation Scale (RASS) | Daily during hospital stay up to 7 days.
  Scores will be charted daily and reviewed in the EMR to determine if differences in sedation are present for patients receiving TEA versus ESPB. The scale ratings range from +4 (combative/violent/immediate danger) to -5 (unarousable).
FiO2 and time on a ventilator | Duration of hospital stay, up to 7 days.
  Will be compared between ESPB and TEA. These values are monitored in the EMR and will be reviewed from the EMR.
Participant satisfaction assessed on a 5 pt. scale | Daily during hospital stay, up to 7 days.
  Assess participant satisfaction of the ESPB and TEA for MRF pain management on a 5 pt scale with 0 being "unsatisfied" and 4 being "very satisfied".
Pain scores | Duration of hospital stay, up to 7 days.
  Pain scores are tracked in the EMR at multiple times during the day. These will be utilized to compare morning and evening charted pain scores to the ones obtained during the morning data collection

CONTACTS AND LOCATIONS:
Overall Officials: Ross Mirman, MD, Principal Investigator — Indiana University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu J, Murphy SL, Kochanek KD, Arias E: Mortality in the United States, 2018. In. Edited by Services USDoHaH. Online: National Center for Health Statistics; 2020.
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Bergeron E, Lavoie A, Clas D, Moore L, Ratte S, Tetreault S, Lemaire J, Martin M. Elderly trauma patients with rib fractures are at greater risk of death and pneumonia. J Trauma. 2003 Mar;54(3):478-85. doi: 10.1097/01.TA.0000037095.83469.4C. PMID 12634526
- [Background] Shorr RM, Crittenden M, Indeck M, Hartunian SL, Rodriguez A. Blunt thoracic trauma. Analysis of 515 patients. Ann Surg. 1987 Aug;206(2):200-5. doi: 10.1097/00000658-198708000-00013. PMID 3606246
- [Background] Moon MR, Luchette FA, Gibson SW, Crews J, Sudarshan G, Hurst JM, Davis K Jr, Johannigman JA, Frame SB, Fischer JE. Prospective, randomized comparison of epidural versus parenteral opioid analgesia in thoracic trauma. Ann Surg. 1999 May;229(5):684-91; discussion 691-2. doi: 10.1097/00000658-199905000-00011. PMID 10235527
- [Background] Govindarajan R, Bakalova T, Michael R, Abadir AR. Epidural buprenorphine in management of pain in multiple rib fractures. Acta Anaesthesiol Scand. 2002 Jul;46(6):660-5. doi: 10.1034/j.1399-6576.2002.460605.x. PMID 12059888
- [Background] Mackersie RC, Karagianes TG, Hoyt DB, Davis JW. Prospective evaluation of epidural and intravenous administration of fentanyl for pain control and restoration of ventilatory function following multiple rib fractures. J Trauma. 1991 Apr;31(4):443-9; discussion 449-51. PMID 1902264
- [Background] Mayberry JC, Trunkey DD. The fractured rib in chest wall trauma. Chest Surg Clin N Am. 1997 May;7(2):239-61. PMID 9156291
- [Background] Karmakar MK, Ho AM. Acute pain management of patients with multiple fractured ribs. J Trauma. 2003 Mar;54(3):615-25. doi: 10.1097/01.TA.0000053197.40145.62. PMID 12634549
- [Background] Cicala RS, Voeller GR, Fox T, Fabian TC, Kudsk K, Mangiante EC. Epidural analgesia in thoracic trauma: effects of lumbar morphine and thoracic bupivacaine on pulmonary function. Crit Care Med. 1990 Feb;18(2):229-31. PMID 2298017
- [Background] Ho AM, Karmakar MK, Critchley LA. Acute pain management of patients with multiple fractured ribs: a focus on regional techniques. Curr Opin Crit Care. 2011 Aug;17(4):323-7. doi: 10.1097/MCC.0b013e328348bf6f. PMID 21716105
- [Background] Gabram SG, Schwartz RJ, Jacobs LM, Lawrence D, Murphy MA, Morrow JS, Hopkins JS, Knauft RF. Clinical management of blunt trauma patients with unilateral rib fractures: a randomized trial. World J Surg. 1995 May-Jun;19(3):388-93. doi: 10.1007/BF00299166. PMID 7638994
- [Background] Jensen CD, Stark JT, Jacobson LL, Powers JM, Joseph MF, Kinsella-Shaw JM, Denegar CR. Improved Outcomes Associated with the Liberal Use of Thoracic Epidural Analgesia in Patients with Rib Fractures. Pain Med. 2017 Sep 1;18(9):1787-1794. doi: 10.1093/pm/pnw199. PMID 27550958
- [Background] De Buck F, Devroe S, Missant C, Van de Velde M. Regional anesthesia outside the operating room: indications and techniques. Curr Opin Anaesthesiol. 2012 Aug;25(4):501-7. doi: 10.1097/ACO.0b013e3283556f58. PMID 22673788
- [Background] Bulger EM, Edwards T, Klotz P, Jurkovich GJ. Epidural analgesia improves outcome after multiple rib fractures. Surgery. 2004 Aug;136(2):426-30. doi: 10.1016/j.surg.2004.05.019. PMID 15300210
- [Background] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Background] Simon BJ, Cushman J, Barraco R, Lane V, Luchette FA, Miglietta M, Roccaforte DJ, Spector R; EAST Practice Management Guidelines Work Group. Pain management guidelines for blunt thoracic trauma. J Trauma. 2005 Nov;59(5):1256-67. doi: 10.1097/01.ta.0000178063.77946.f5. No abstract available. PMID 16385313
- [Background] Geerts WH, Jay RM, Code KI, Chen E, Szalai JP, Saibil EA, Hamilton PA. A comparison of low-dose heparin with low-molecular-weight heparin as prophylaxis against venous thromboembolism after major trauma. N Engl J Med. 1996 Sep 5;335(10):701-7. doi: 10.1056/NEJM199609053351003. PMID 8703169
- [Background] Rogers FB, Cipolle MD, Velmahos G, Rozycki G, Luchette FA. Practice management guidelines for the prevention of venous thromboembolism in trauma patients: the EAST practice management guidelines work group. J Trauma. 2002 Jul;53(1):142-64. doi: 10.1097/00005373-200207000-00032. No abstract available. PMID 12131409
- [Background] Malekpour M, Hashmi A, Dove J, Torres D, Wild J. Analgesic Choice in Management of Rib Fractures: Paravertebral Block or Epidural Analgesia? Anesth Analg. 2017 Jun;124(6):1906-1911. doi: 10.1213/ANE.0000000000002113. PMID 28525509
- [Background] Mohta M, Verma P, Saxena AK, Sethi AK, Tyagi A, Girotra G. Prospective, randomized comparison of continuous thoracic epidural and thoracic paravertebral infusion in patients with unilateral multiple fractured ribs--a pilot study. J Trauma. 2009 Apr;66(4):1096-101. doi: 10.1097/TA.0b013e318166d76d. PMID 19359920
- [Background] Osinowo OA, Zahrani M, Softah A. Effect of intercostal nerve block with 0.5% bupivacaine on peak expiratory flow rate and arterial oxygen saturation in rib fractures. J Trauma. 2004 Feb;56(2):345-7. doi: 10.1097/01.TA.0000046257.70194.2D. PMID 14960978
- [Background] Short K, Scheeres D, Mlakar J, Dean R. Evaluation of intrapleural analgesia in the management of blunt traumatic chest wall pain: a clinical trial. Am Surg. 1996 Jun;62(6):488-93. PMID 8651535
- [Background] Lonnqvist PA, MacKenzie J, Soni AK, Conacher ID. Paravertebral blockade. Failure rate and complications. Anaesthesia. 1995 Sep;50(9):813-5. doi: 10.1111/j.1365-2044.1995.tb06148.x. PMID 7573876
- [Background] Richardson J, Sabanathan S, Mearns AJ, Shah RD, Goulden C. A prospective, randomized comparison of interpleural and paravertebral analgesia in thoracic surgery. Br J Anaesth. 1995 Oct;75(4):405-8. doi: 10.1093/bja/75.4.405. PMID 7488477
- [Background] Shanti CM, Carlin AM, Tyburski JG. Incidence of pneumothorax from intercostal nerve block for analgesia in rib fractures. J Trauma. 2001 Sep;51(3):536-9. doi: 10.1097/00005373-200109000-00019. PMID 11535906
- [Background] Kunhabdulla NP, Agarwal A, Gaur A, Gautam SK, Gupta R, Agarwal A. Serratus anterior plane block for multiple rib fractures. Pain Physician. 2014 Sep-Oct;17(5):E651-3. No abstract available. PMID 25247916
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Jain K, Jaiswal V, Puri A. Erector spinae plane block: Relatively new block on horizon with a wide spectrum of application - A case series. Indian J Anaesth. 2018 Oct;62(10):809-813. doi: 10.4103/ija.IJA_263_18. PMID 30443066
- [Background] Adhikary SD, Pruett A, Forero M, Thiruvenkatarajan V. Erector spinae plane block as an alternative to epidural analgesia for post-operative analgesia following video-assisted thoracoscopic surgery: A case study and a literature review on the spread of local anaesthetic in the erector spinae plane. Indian J Anaesth. 2018 Jan;62(1):75-78. doi: 10.4103/ija.IJA_693_17. PMID 29416155
- [Background] Barrios A, Camelo J, Gomez J, Forero M, Peng PWH, Visbal K, Cadavid A. Evaluation of Sensory Mapping of Erector Spinae Plane Block. Pain Physician. 2020 Jun;23(3):E289-E296. PMID 32517405
- [Background] El-Boghdadly K, Pawa A. The erector spinae plane block: plane and simple. Anaesthesia. 2017 Apr;72(4):434-438. doi: 10.1111/anae.13830. Epub 2017 Feb 11. No abstract available. PMID 28188611
- [Background] Shibata Y, Kampitak W, Tansatit T. The Novel Costotransverse Foramen Block Technique: Distribution Characteristics of Injectate Compared with Erector Spinae Plane Block. Pain Physician. 2020 Jun;23(3):E305-E314. PMID 32517407
- [Background] Nandhakumar A, Nair A, Bharath VK, Kalingarayar S, Ramaswamy BP, Dhatchinamoorthi D. Erector spinae plane block may aid weaning from mechanical ventilation in patients with multiple rib fractures: Case report of two cases. Indian J Anaesth. 2018 Feb;62(2):139-141. doi: 10.4103/ija.IJA_599_17. PMID 29491521
- [Background] Yayik AM, Ahiskalioglu A, Celik EC, Ay A, Ozenoglu A. [Continuous erector spinae plane block for postoperative analgesia of multiple rib fracture surgery: case report]. Braz J Anesthesiol. 2019 Jan-Feb;69(1):91-94. doi: 10.1016/j.bjan.2018.08.001. Epub 2018 Nov 2. PMID 30392675
- [Background] Cao J, Gao X, Zhang X, Li J, Zhang J. Feasibility of laryngeal mask anesthesia combined with nerve block in adult patients undergoing internal fixation of rib fractures: a prospective observational study. BMC Anesthesiol. 2020 Jul 15;20(1):170. doi: 10.1186/s12871-020-01082-y. PMID 32669087
- [Background] Adhikary SD, Liu WM, Fuller E, Cruz-Eng H, Chin KJ. The effect of erector spinae plane block on respiratory and analgesic outcomes in multiple rib fractures: a retrospective cohort study. Anaesthesia. 2019 May;74(5):585-593. doi: 10.1111/anae.14579. Epub 2019 Feb 10. PMID 30740657
- [Background] Gursoy C, Kuscu Y, Demirbilek SG. Pain Management for Traumatic Rib Fractures with ESP Block in ICU. J Coll Physicians Surg Pak. 2020 Mar;30(3):318-320. doi: 10.29271/jcpsp.2020.03.318. PMID 32169144
- [Background] Liu R, Clark L, Bautista A. Unilateral Bilevel Erector Spinae Plane Catheters for Flail Chest: A Case Report. A A Pract. 2020 May;14(7):e01211. doi: 10.1213/XAA.0000000000001211. PMID 32371819
- [Background] Epidural Anesthesia and Analgesia [https://www.nysora.com/regional-anesthesia-for-specific-surgical-procedures/abdomen/epidural-anesthesia-analgesia/]
- [Background] Bomberg H, Bayer I, Wagenpfeil S, Kessler P, Wulf H, Standl T, Gottschalk A, Doffert J, Hering W, Birnbaum J, Spies C, Kutter B, Winckelmann J, Liebl-Biereige S, Meissner W, Vicent O, Koch T, Sessler DI, Volk T, Raddatz A. Prolonged Catheter Use and Infection in Regional Anesthesia: A Retrospective Registry Analysis. Anesthesiology. 2018 Apr;128(4):764-773. doi: 10.1097/ALN.0000000000002105. PMID 29420315